CLINICAL TRIAL: NCT02904473
Title: Goals for Reaching Optimum Wellness (GROWell): A Pilot Study of a Dietary Intervention During Pregnancy
Brief Title: Goals for Reaching Optimum Wellness (GROWell)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00071547
Record Dates: First submitted 2016-08-31; First posted 2016-09-19 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2018-10

CONDITIONS: Pregnant Women

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- GROWell (Experimental): GROWell incorporates 4 elements: phone coaching, goal setting, self-monitoring of behavior and skills training. These interactions take place on a study subject's cell phone, through text messaging, and phone calls with a dietician coach. At study initiation, the subject takes a short survey, after which the intervention algorithm assigns up to 4 tailored behavior change goals from the GROWell library. Goals are tailored to the subject's needs as indicated by the initial survey. Subjects self-monitor adherence weekly via text, responding to prompts from the system regarding their level of success with a given goal. Via text they receive immediate tailored feedback regarding their current adherence and long-term progress.
  Interventions: Other: GROWell
- Attention Support Control (ASC) (No Intervention): The ASC control arm of the study involves one coaching call at baseline, regarding prenatal diet. Weekly text or IVR messages will focus on pregnancy, labor, delivery, and early infancy education.
- Usual Care (USC) (No Intervention): The USC will receive no intervention. They will simply complete baseline and follow-up CASI and blood draw.

INTERVENTIONS:
Other: GROWell — The GROWell intervention is a mobile health technology, including diet tracking, skills training and tailored feedback based on digital and human support strategies. Its message content is geared toward healthy diet change during pregnancy.
  Arms: GROWell

SUMMARY:
This is a pilot study to assess the feasibility, acceptability and preliminary efficacy of the GROWell diet intervention. The objective of this study is to determine whether the GROWell intervention can help transition women from consuming a Western diet to consuming a prudent diet (characterized by consumption of primarily fruits, vegetables, healthy fats, lean proteins, and whole grains) during pregnancy. Efficacy will be measured as change in dietary components, using a Food Frequency Questionnaire (FFQ) at baseline and at a follow up visit at 37 weeks gestation.

The GROWell intervention is a mobile health technology that uses interactive text messaging and dietician coaching calls, and may be effective in transitioning pregnant women from a Western to a prudent diet during an approximately 6 month intervention period. GROWell results will be measured against an Attention Support Control (ASC) arm, where participants will receive messaging that is pregnancy rather than diet focused, and a Usual Care (USC) arm, where participants will not receive text messages or study coaching.

Results from this study will be used to support a grant submission for a larger study, aiming to investigate the GROWell intervention and prudent diet consumption as preventatives against postpartum depression.

DETAILED DESCRIPTION:
The GROWell intervention is a mobile health technology, including diet tracking, skills training and tailored feedback based on digital and human support strategies. Its structure is based on the iOTA (interactive obesity treatment approach), designed for dietary change, obesity, and chronic disease management, with message content modified for healthy diet change during pregnancy.

GROWell incorporates 4 elements: phone coaching, goal setting, self-monitoring of behavior and skills training. These interactions take place on a study subject's cell phone, through text messaging, and phone calls with a dietician coach. At the initiation of the intervention, the subject takes a short survey, after which the intervention algorithm assigns up to 4 tailored behavior change goals from the GROWell library. Examples of goals would be to eliminate fast food from the diet, or to limit red meat. Goals are tailored to the subject's needs as indicated by the initial survey, so if for example the subject doesn't eat fast food, that goal is not assigned. The algorithm prioritizes behaviors in highest need of change, and those for which participant has high self-efficacy and readiness based on the survey responses. Subjects self-monitor adherence weekly via text, responding to prompts from the system regarding their level of success with a given goal. Via text they receive immediate tailored feedback regarding their current adherence and long-term progress.

Feedback includes showing progress trends, reinforcing success, and offering motivational strategies to support behavior change based on the self-monitoring data. To support the next week's efforts, the algorithm tailors feedback, selecting content from a skills training library and sending materials to assist behavior change efforts. Skills training materials include online handouts, featuring content that discusses the adoption of healthy dietary changes in pregnancy. A set of skills training materials exists for each goal in the library. When a subject is assigned a goal, they receive a link to the training materials for that goal over the phone.

The human support component of the intervention relies in part on the GROWell platform's interface, which allows diet coaches to view participant data. This information is then used to inform feedback during coaching calls. These 15-minute conversations will be guided by principles of motivational interviewing (MI). In each session, the dietician coach and the subject will discuss self-monitoring data and reinforce its importance, discuss barrier reduction strategies and skills training content, and engaging community resources. The GROWell study will implement a series of dietician coaching calls starting weekly for the first month and decreasing in frequency to biweekly during the study period, totaling approximately 12 calls depending on delivery date.

The ASC control arm of the study involves more limited intervention. There will be one coaching call at baseline, regarding prenatal diet. Weekly text or IVR messages will focus on pregnancy, labor, delivery, and early infancy education.

The USC will receive no intervention. They will simply complete baseline and follow-up questionnaires.

Participants on all arms may opt to have blood drawn at the baseline visit and the follow up visit for an optional biomarker study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 44
* Read and understand English
* Receiving prenatal care at Duke Medicine
* Prepregnancy BMI ≥25 and <35
* Within 14 to <20 weeks gestation
* Singleton, uncomplicated pregnancy [no preexisting diabetes, hypertension, etc.]
* Non-smoking for at least 6 months
* Nulliparous, or >24 months since previous pregnancy
* No current depression as documented in the medical record
* Has a cell phone with texting capability [smartphone not required], and is willing to use it at their expense for study purposes

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of the GROWell intervention | 37 Weeks Gestation
  Feasibility will be assessed based on the number and percent of women enrolled vs. approached, vs. completing all study assessments.
Acceptability of the GROWell intervention | 37 Weeks Gestation
  Acceptability measures are participant adherence to digital communications and coaching calls. Subjects will also rate the intervention regarding perceived helpfulness, relationship with their coach, etc.
Efficacy- change in dietary components from Baseline to 37 Weeks Gestation | Baseline to 37 Weeks Gestation
  Efficacy will be measured as change in dietary components between the arms, as reported in a Food Frequency Questionnaire (FFQ) reflecting Western or prudent intake over the intervention period. Switching from a Western to a prudent diet is defined as consuming a prudent diet on most days, as determined by questionnaire responses.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Ann Simmons, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States